CLINICAL TRIAL: NCT06930339
Title: Portable Neuromodulation Stimulator Registry for People With Multiple Sclerosis
Acronym: PoNSREM
Status: Active, not recruiting | Type: Observational
Sponsor: Helius Medical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: HMI-MS-PoNS-RE001
Record Dates: First submitted 2025-03-25; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis
Keywords: Gait deficit, PoNS
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Portable Neuromodulation Stimulator (PoNS) — No intervention

SUMMARY:
The Registry will be designed to gather information over 3 years. This important health economic information will help to establish the value of the PoNS Device on key therapeutic outcomes. These outcomes will include:

disease-associated injury risks (i.e., falls), onset of new comorbidities and/or worsening/improvement of existing medical condition(s) (other than gait deficit/impairment), need for new pharmacological/non-pharmacological intervention or increase/decrease of ongoing pharmacotherapy or other non-pharmacological intervention, increase/decrease of in patient/outpatient hospital and/or office visits or stays, side effects.

By participation in the Registry, patients and physicians will be providing Helius with access to information about medical history, medical diagnoses, clinical symptom presentations, vocational information, medications, pharmacologic and non-pharmacologic prescriptions, hospitalization and healthcare visits, and any reported therapy's adverse events.

ELIGIBILITY:
Inclusion Criteria: none

* Diagnosis of gait deficit due to MS

Exclusion Criteria: none

* unable to ambulate with or without an assisting device

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry is designed to collect retrospective clinical/medical outcome data on the therapeutic response of MS patients with gait deficit who underwent at least an initial 14-week PoNS Therapy course.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of PoNS Therapy as measured by self-reported change in symptomatology | 3 years
  Balance and Gait deficit improvement after physical therapy rehabilitation with PoNS device over one or more courses of 14-week therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Helius Medical, Newtown, Pennsylvania, United States